CLINICAL TRIAL: NCT03016221
Title: Local Changes of Skin Characteristics During and After an Application of a Topical Product With a Warming or Cooling Effect - a Randomized, Controlled Clinical Trial
Brief Title: Local Changes of Skin Characteristics After an Application of a Topical Product With a Warming or Cooling Effect
Acronym: SRPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2016-01541
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: local skin responses; hyperemia; thermal sensation; topical warming ointments; topical cooling ointments; skin perfusion; subjective thermal sensation; muscle tissue oxygenation; skin temperature; skin redness; erythema
MeSH Terms: conditions — Hyperemia; Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Axanova hot gel (Experimental): Intervention: Axanova hot gel is a topical product with a warming effect. In a single application 3g of the product is applied in an area of 10cm x 10cm on the unilateral lumbar back until it has been completely absorbed by the skin.
  Interventions: Other: Axanova hot gel
- Axanova hot gel control (No Intervention): No product application. The contralateral lumbar back side acts as a Axanova hot gel control.
- Axanova activ gel (Experimental): Intervention: Axanova activ gel is a topical product with a revulsive effect. In a single application 3g of the product is applied in an area of 10cm x 10cm on the unilateral lumbar back until it has been completely absorbed by the skin.
  Interventions: Other: Axanova activ gel
- Axanova activ gel control (No Intervention): No product application. The contralateral lumbar back side acts as a Axanova activ gel control.
- Perskindol Dolo Gel (Experimental): Intervention: Perskindol Dolo Gel is a topical product with a warming effect. In a single application 3g of the product is applied in an area of 10cm x 10cm on the unilateral lumbar back until it has been completely absorbed by the skin.
  Interventions: Other: Perskindol Dolo Gel
- Perskindol Dolo Gel control (No Intervention): No product application. The contralateral lumbar back side acts as a Perskindol Dolo Gel control.
- Perskindol Classic Gel (Experimental): Intervention: Perskindol Classic Gel is a topical product with a revulsive effect. In a single application 3g of the product is applied in an area of 10cm x 10cm on the unilateral lumbar back until it has been completely absorbed by the skin.
  Interventions: Other: Perskindol Classic Gel
- Perskindol Classic Gel control (No Intervention): No product application. The contralateral lumbar back side acts as a Perskindol Classic Gel control.
- Perskindol Cool Kühl-Gel (Experimental): Intervention: Perskindol Cool Kühl-Gel is a topical product with a cooling effect. In a single application 3g of the product is applied in an area of 10cm x 10cm on the unilateral lumbar back until it has been completely absorbed by the skin.
  Interventions: Other: Perskindol Cool Kühl-Gel
- Perskindol Cool Kühl-Gel control (No Intervention): No product application. The contralateral lumbar back side acts as a Perskindol Cool Kühl-Gel control.
- Dolor-X Hot Gel (Experimental): Intervention: Dolor-X Hot Gel is a topical product with a warming effect. In a single application 3g of the product is applied in an area of 10cm x 10cm on the unilateral lumbar back until it has been completely absorbed by the skin.
  Interventions: Other: Dolor-X Hot Gel
- Dolor-X Hot Gel control (No Intervention): No product application. The contralateral lumbar back side acts as a Dolor-X Hot Gel control.
- Dolor-X Classic Gel (Experimental): Intervention: Dolor-X Classic Gel is a topical product with a revulsive effect. In a single application 3g of the product is applied in an area of 10cm x 10cm on the unilateral lumbar back until it has been completely absorbed by the skin.
  Interventions: Other: Dolor-X Classic Gel
- Dolor-X Classic Gel control (No Intervention): No product application. The contralateral lumbar back side acts as a Dolor-X Classic Gel control.
- Dolor-X Cool Gel (Experimental): Intervention: Dolor-X Cool Gel is a topical product with a cooling effect. In a single application 3g of the product is applied in an area of 10cm x 10cm on the unilateral lumbar back until it has been completely absorbed by the skin.
  Interventions: Other: Dolor-X Cool Gel
- Dolor-X Cool Gel control (No Intervention): No product application. The contralateral lumbar back side acts as a Dolor-X Cool Gel control.

INTERVENTIONS:
Other: Axanova hot gel — Axanova hot gel is a topical product with a warming effect. It contains menthol, pine needle oil, wintergreen oil, rosemary oil, eucalyptus oil, incense oil.
  Arms: Axanova hot gel
Other: Axanova activ gel — Axanova activ gel is a topical product with a revulsive effect. It contains menthol, pine needle oil, orange oil, lemon oil, wintergreen oil, glycosaminoglycans.
  Arms: Axanova activ gel
Other: Perskindol Dolo Gel — Perskindol Dolo Gel is a topical product with a warming effect. It contains wintergreen oil, pine needle oil, aromatics, excipients.
  Arms: Perskindol Dolo Gel
Other: Perskindol Classic Gel — Perskindol Classic Gel is a topical product with a revulsive effect. It contains menthol, wintergreen oil, pine needle oil, lemon oil, orange peel oil, lemon bergamot oil, rosemary oil, lavender oil, excipients.
  Arms: Perskindol Classic Gel
Other: Perskindol Cool Kühl-Gel — Perskindol Cool Kühl-Gel is a topical product with a cooling effect. It contains levomenthol, color E131, aromatics, excipients.
  Arms: Perskindol Cool Kühl-Gel
Other: Dolor-X Hot Gel — Dolor-X Hot Gel is a topical product with a warming effect. It contains isopropyl alcohol, water, menthol, hyprolose, camphor, trometamol, paprika, wintergreen oil, excipients.
  Arms: Dolor-X Hot Gel
Other: Dolor-X Classic Gel — Dolor-X Classic Gel is a revulsive product. It contains water, isopropyl alcohol, menthol, spruce, hyprolose, trometamol, wintergreen oil, excipients.
  Arms: Dolor-X Classic Gel
Other: Dolor-X Cool Gel — Dolor-X Cool Gel is a cooling product. It contains water, isopropyl alcohol, menthol, trometamol, color E131, excipients.
  Arms: Dolor-X Cool Gel

SUMMARY:
The use of topical over-the-counter (OTC) products with a warming or cooling effect is widespread in the fields of sport, physiotherapy and in private households. Advertisements for such products promise pain relief when suffering from musculoskeletal disorders such as muscle tension, rheumatism or acute injuries, e.g. sprains. In literature, there are only little information about the efficacy and the physiological mechanisms of topical warming or cooling products. Therefore, the aim of this study is to investigate the local skin characteristics during and after an application of a topical product with a warming or cooling effect.

DETAILED DESCRIPTION:
The use of topical products for local pain relief in chronic or acute musculoskeletal disorders is widely used. Despite the widespread use of these products, there is missing information on the physiological mechanisms and efficacy of topical warming and cooling ointments. Most of the existing literature is about the efficacy of topical non-steroidal anti-inflammatory drug (NSAID)-products on chronic pain in osteoarthritis. Furthermore, one study tested the cooling effect of gels with different menthol concentrations. They found that, regardless of the concentration, the skin temperature was reduced up to one hour post application in the area of application.

The aim of our study is to evaluate the change of skin characteristics after a single application of a warming or cooling topical product on healthy subjects. Outcome parameters include skin perfusion, temperature, skin redness and subjective thermal sensation. We only selected products in form of alcohol based ointments, menthol or wintergreen oil. Sprays and patches were excluded.

The application area is the unilateral lumbar back region, whereas the contralateral side serves as control area. After an acclimatization period, baseline measurements are performed, followed by standardized application of the topical product. The local skin responses are measured in 10 mins time increments up to one hour.

ELIGIBILITY:
Inclusion Criteria:

* no existing musculoskeletal disorders in the region of interest
* no surgery in the region of interest in the last year
* healthy skin conditions in the region of interest

Exclusion Criteria:

* fear of treatment
* regular intake of drugs, excluding contraceptives
* metal implants in the region between C7 and sacrum, including hip joints
* lack of epicritic and protopathic skin sensitivity
* renal insufficiency
* bronchial asthma
* pregnancy/lactation
* type 1 or 2 diabetes mellitus
* polyneuropathy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
local skin perfusion | during one hour post application
  local skin perfusion will be measured with a laser speckle instrument
local skin redness | during one hour post application
  local skin redness (erythema) will be measured with a chromameter
skin surface temperature | during one hour post application
  skin surface temperature will be measured with thermochrons, infrared thermometer and thermal imaging camera
local muscle tissue oxygenation | during one hour post application
  local muscle tissue oxygenation will be measured with near infrared spectroscopy
subjective temperature sensation | during one hour post application
  subjective temperature sensation will be evaluated with a thermal comfort questionnaire

SECONDARY OUTCOMES:
skin perfusion directly next to the application area | during one hour post application
  skin perfusion will be measured with a laser speckle instrument
skin redness directly next to the application area | during one hour post application
  skin redness (erythema) will be measured with a chromameter
skin temperature directly next to the application area | during one hour post application
  skin surface temperature will be measured with thermochrons, infrared thermometer and thermal imaging camera
muscle tissue oxygenation directly next to the application area | during one hour post application
  muscle tissue oxygenation will be measured with near infrared spectroscopy
subjective temperature sensation directly next to the application area | during one hour post application
  subjective temperature sensation will be evaluated with a thermal comfort questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- SUPSI, Landquart, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No